CLINICAL TRIAL: NCT01770769
Title: Undisplaced Femoral Neck Fractures in Patients Aged 70 Years and Older: A Multicentre Randomised Controlled Trial Comparing Internal Fixation to Hemiarthroplasty
Brief Title: Undisplaced Femoral Neck Fractures in the Elderly: A Trial Comparing Internal Fixation to Hemiarthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Akershus (Other)
Collaborators: University of Oslo (Other); Asker & Baerum Hospital (Other); Sykehuset Innlandet HF (Other); Vestre Viken Hospital Trust (Other)
Responsible Party: Principal Investigator, Filip C Dolatowski, Principal Investigator, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEM-2011/2296
Record Dates: First submitted 2012-04-25; First posted 2013-01-18 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Femoral Neck Fractures
Keywords: Femoral Neck Fracture; undisplaced; minimally displaced; internal fixation; hemiarthroplasty; harris hip score; hospital cost; society cost; quality of life; Timed Up and go test
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Hemiarthroplasty; Fracture Fixation, Internal

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Internal fixation - standard treatment (Active Comparator): Internal fixation with two parallel cancellous screws (Hip Pins(R)) Current standard treatment
  Interventions: Device: internal fixation
- Hemi - arthroplasty (Experimental): cemented Hemi - arthroplasty (Exeter(R)) modular system V40 by Stryker. Refobacin cement.
  Interventions: Device: Hemi - arthroplasty

INTERVENTIONS:
Device: Hemi - arthroplasty — modular hemiarthroplasty
  Other Names: Hemiarthroplasty by Stryker - Exeter V40(R); Hemiarthroplasty by DePuy - Corail; Refobacin® Bone Cement R & Biomet; Cloxacillin or cephalothin perioperative prophylaxis; Fragmin (Dalteparin) anticoagulation for 2 wks
  Arms: Hemi - arthroplasty
Device: internal fixation — Two cancellous parallel screws - internal fixation of the femoral neck fracture
  Other Names: Hip Pins (R); Cloxacillin or cephalothin perioperative prophylaxis; Fragmin (Dalteparin) anticoagulation for 2 wks
  Arms: Internal fixation - standard treatment

SUMMARY:
Clinical research during the last ten years has revealed that elderly patients with a displaced femoral neck fracture should be treated with arthroplasty instead of closed reduction of the fracture followed by internal fixation with pins or screws. Few clinical trials have addressed undisplaced or minimally displaced fractures of the femoral neck. These fractures have been associated with a good prognosis and likewise a good functional outcome. However, recent articles present far less favorable results, with high re-operation rates (10-15%), reduced function, and pain on walking after internal fixation. Indirect comparing studies, suggest that hemiarthroplasty may yield better functional outcomes and lower re-operation rates. Approximately 20% of all femoral neck fractures in patients aged 70 years or older are minimally displaced or undisplaced. Hence the investigators call for a randomised controlled trial comparing pain, function, walking ability, quality of life, re-operation rates and complications after internal fixation versus hemiarthroplasty in patients aged 70 years and older.

DETAILED DESCRIPTION:
The consequences of a femoral neck fracture still have a substantial impact on the individual patient´s health as well as on society. Approximately 5000 individuals suffer a fracture of the femoral neck annually in Norway. The mortality rate approximates 25% during the first year after this injury. The hospital costs of treating a single femoral neck fracture, have been estimated to 20 000 euros.

In spite of relatively well-documented treatment protocols, there is still a need for prospective randomised controlled trials to determine the optimal treatment of certain sub-groups of patients presenting with a femoral neck fracture.

Several studies with a high level of evidence have elucidated management of displaced femoral neck fractures. There is increasing evidence favouring joint replacement surgery over internal fixation when treating displaced femoral neck fractures. However, management of undisplaced and minimally displaced femoral neck fractures has received less attention.

According to the Cochrane Library, there are no randomised controlled trials comparing internal fixation to hemiarthroplasty in patients with undisplaced femoral neck fractures. Previous studies have focused mostly on fracture healing, equating fracture union and success. However, recent studies report decreased functional and life quality scores amongst patients with undisplaced femoral neck fractures treated with internal fixation. The control group in these studies consists of patients with a displaced femoral neck fracture treated with hemi - arthroplasty. Zlowodzki et al showed, by means of validated assessment scores, that patients with internally fixated undisplaced femoral neck fractures often experience shortening of the injured limb. Then again, this is associated with lower functional and life quality scores. In Rogmark´s series of patients with undisplaced femoral neck fractures treated with internal fixation, 25% patients report daily pain from the affected hip upon walking, one and a half year after surgery. Gjertsen et al analysed data for the Norwegian hip fracture registry from more than 4000 patients to demonstrate that treatment with hemiarthroplasty, due to a displaced femoral neck fracture, is associated with better function and less pain than treatment with internal fixation due to an undisplaced femoral neck fracture.

Thus, our research group will conduct a prospective randomised controlled trial to identify any differences in clinical outcome after surgical treatment of undisplaced femoral neck fractures in patients aged 70 years and older. The two methods that will be compared are internal fixation with two screws and modern modular hemiarthroplasty. The primary outcome measure is a difference of at least 10 points in Harris Hip Score (95% power, standard deviation approximates 15 points from previous Norwegian patient series). The primary follow-up length is set to two years, but a long-term follow-up five years after surgery is also planned. It is important to include the cognitively impaired patients as they account for 20-25% of the study population. Patients who cannot provide informed consent due to impaired cognitive function, are included if consent is provided by a family member or relative.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 years or older
* Undisplaced or minimally displaced intracapsular femoral neck fracture (Garden I/II)
* Patient able to walk before injury (all aids allowed)
* Patient lives within the catchment area of the three involved centres

Exclusion Criteria:

* Displaced fractures (Garden III/IV) and impacted fractures with minimal varus
* Pathologic fracture
* Current soft tissue or deep infection in the hip or pelvis area
* ASA IV patients as classified by the anesthesiologist on call
* Other contraindications to either of the two methods compared
* Temporarily impaired cognitive function:

(That is when the patient is judged as unable to provide an informed consent by the surgeon on call and there is no previous history of impaired cognitive function as documented by previous hospital record or a family member / proxy)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 220 (Actual)
Dates: Start 2012-02-06 (Actual); Primary Completion 2020-02-06 (Estimated); Study Completion 2020-02-06 (Estimated)

PRIMARY OUTCOMES:
Change in Harris Hip Score of 10 points or more. | Baseline prior to fracture, 3 months, 1 year and 2 years
  Harris hip score - a validated outcome measure to evaluate hip fracture intervention The physiotherapist recording the Harris Hips Score after 3 months, 1 year and two years is blinded. Clinical examination of the hip is carried out with masking of proximal thigh by proper clothes.

SECONDARY OUTCOMES:
Euro-Quol 5 dimension (Eq5d) | Baseline prior to fracture, 3 months, 1 year and 2 years
  Eq5D a validated measure of quality of life and to be utilised in health economic models comparing hospital and society costs of the two surgical methods compared. The investigator is blinded.
Numeric pain intensity scale (0-10) | Two weeks prior to fracture (retrospective), at discharge at an average 3-5 days after surgery, after 3 months, 1 year and 2 years
  Visual analog scale variant with numbers from ranging from zero (no pain) to ten (worst possible pain). The investigator is blinded.
Timed Up and Go test (TUG test) | 3 months, 1 year and 2 years
  Patient sits on a chair, rises, walks 3 meters passing a mark, turns around, walks back and sits down. The time is recorded in seconds. The investigator is blinded.
Reoperation rate | 5 years after surgery
  All complications are continually recorded in both trial arms.
Death | 5 years after surgery
  All deaths are recorded
Mini mental state(MMSE-NR) | 3 months
  Mini mental state is recorded only at 3 months follow-up
Hospital and society costs | at baseline prior to fracture, at discharge, 3 months, 1 year and 2 years
  Use of governmental and private health care services and assistance by family members and relatives are all recorded. Validated health economical models are used to calculate the costs.

CONTACTS AND LOCATIONS:
Overall Officials: Torbjørn Omland, Professor, Study Chair — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lillestrøm, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Data planned published in English in a peer-reviewed medical journal

REFERENCES:
- [Background] Gjertsen JE, Fevang JM, Matre K, Vinje T, Engesaeter LB. Clinical outcome after undisplaced femoral neck fractures. Acta Orthop. 2011 Jun;82(3):268-74. doi: 10.3109/17453674.2011.588857. PMID 21619501
- [Background] Parker MJ, Gurusamy K. Internal fixation versus arthroplasty for intracapsular proximal femoral fractures in adults. Cochrane Database Syst Rev. 2006 Oct 18;2006(4):CD001708. doi: 10.1002/14651858.CD001708.pub2. PMID 17054139
- [Background] Frihagen F, Waaler GM, Madsen JE, Nordsletten L, Aspaas S, Aas E. The cost of hemiarthroplasty compared to that of internal fixation for femoral neck fractures. 2-year results involving 222 patients based on a randomized controlled trial. Acta Orthop. 2010 Aug;81(4):446-52. doi: 10.3109/17453674.2010.492763. PMID 20515432
- [Background] Heetveld MJ, Rogmark C, Frihagen F, Keating J. Internal fixation versus arthroplasty for displaced femoral neck fractures: what is the evidence? J Orthop Trauma. 2009 Jul;23(6):395-402. doi: 10.1097/BOT.0b013e318176147d. PMID 19550224
- [Background] Frihagen F, Nordsletten L, Madsen JE. Hemiarthroplasty or internal fixation for intracapsular displaced femoral neck fractures: randomised controlled trial. BMJ. 2007 Dec 15;335(7632):1251-4. doi: 10.1136/bmj.39399.456551.25. Epub 2007 Dec 4. PMID 18056740
- [Background] Rogmark C, Carlsson A, Johnell O, Sernbo I. A prospective randomised trial of internal fixation versus arthroplasty for displaced fractures of the neck of the femur. Functional outcome for 450 patients at two years. J Bone Joint Surg Br. 2002 Mar;84(2):183-8. doi: 10.1302/0301-620x.84b2.11923. PMID 11922358
- [Background] Bjorgul K, Reikeras O. Hemiarthroplasty in worst cases is better than internal fixation in best cases of displaced femoral neck fractures: a prospective study of 683 patients treated with hemiarthroplasty or internal fixation. Acta Orthop. 2006 Jun;77(3):368-74. doi: 10.1080/17453670610046271. PMID 16819673
- [Background] Rogmark C, Flensburg L, Fredin H. Undisplaced femoral neck fractures--no problems? A consecutive study of 224 patients treated with internal fixation. Injury. 2009 Mar;40(3):274-6. doi: 10.1016/j.injury.2008.05.023. Epub 2008 Dec 13. PMID 19070851
- [Background] Zlowodzki M, Ayeni O, Petrisor BA, Bhandari M. Femoral neck shortening after fracture fixation with multiple cancellous screws: incidence and effect on function. J Trauma. 2008 Jan;64(1):163-9. doi: 10.1097/01.ta.0000241143.71274.63. PMID 18188116
- [Background] Zlowodzki M, Brink O, Switzer J, Wingerter S, Woodall J Jr, Petrisor BA, Kregor PJ, Bruinsma DR, Bhandari M. The effect of shortening and varus collapse of the femoral neck on function after fixation of intracapsular fracture of the hip: a multi-centre cohort study. J Bone Joint Surg Br. 2008 Nov;90(11):1487-94. doi: 10.1302/0301-620X.90B11.20582. PMID 18978271
- [Background] Zlowodzki M, Jonsson A, Paulke R, Kregor PJ, Bhandari M. Shortening after femoral neck fracture fixation: is there a solution? Clin Orthop Relat Res. 2007 Aug;461:213-8. doi: 10.1097/BLO.0b013e31805b7ec4. PMID 17415006
- [Background] Frihagen F, Grotle M, Madsen JE, Wyller TB, Mowinckel P, Nordsletten L. Outcome after femoral neck fractures: a comparison of Harris Hip Score, Eq-5d and Barthel Index. Injury. 2008 Oct;39(10):1147-56. doi: 10.1016/j.injury.2008.03.027. Epub 2008 Jul 25. PMID 18656868